CLINICAL TRIAL: NCT00936065
Title: A Multicenter, Randomized, Open Pilot Trial Assessing the Efficacy and Safety of Etanercept 50 mg Twice Weekly Followed Etanercept 25mg Twice Weekly, the Combination of Etanercept 25 mg Twice Weekly and Acitretin and Acitretin Alone in Patients With Moderate to Severe Psoriasis
Brief Title: Study Evaluating the Efficacy and Safety of Etanercept and Acitretin in Korean Patient With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A6-4625; B1801065
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-03

CONDITIONS: Moderate to Severe Psoriasis
Keywords: Etanercept; Acitretin; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept; Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator)
  Interventions: Drug: Etanercept
- Group B (Experimental)
  Interventions: Drug: Etanercept + Acitretin
- Group C (Active Comparator)
  Interventions: Drug: Acitretin

INTERVENTIONS:
Drug: Etanercept — Etanercept at a dose of 50mg twice weekly for 12 weeks followed by 25mg twice weekly for 12 weeks
  Other Names: Etanercept 50mg followed by 25mg
  Arms: Group A
Drug: Etanercept + Acitretin — Combination of etanercept at a dose of 25mg twice weekly and acitretin 10mg BID for 24 weeks
  Other Names: Etancercept 25mg and Acitretin 10mg
  Arms: Group B
Drug: Acitretin — Acitretin at a dose of 10mg BID for 24 weeks
  Other Names: Acitretin 10mg
  Arms: Group C

SUMMARY:
To compare the efficacy of ETN 50mg twice weekly for 12 weeks followed by reduction to a maintenance dose of 25mg twice weekly at week 24 with that of combination of ETN 25 mg Twice Weekly plus Acitretin 10mg BID at week 24 in subjects with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Active, moderate to severe psoriasis defined by the following criteria: Clinically stable, plaque psoriasis involving more than 10% body surface area (BSA) or PASI 10.
* In the opinion of the investigator, failure, intolerance, contraindication or not a candidate for the following: Methotrexate (MTX), cyclosporine, and psoralen plus ultraviolet A radiation (PUVA) therapy.
* Negative urine pregnancy test before the first dose of study drug in all female patients

Exclusion Criteria:

* Evidence of skin conditions (e.g., eczema) other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis.
* Any rheumatologic disease such as rheumatoid arthritis, psoriatic arthritis, gout, systemic lupus erythematous, systemic vasculitis, scleroderma and polymyositis, or associated syndromes.
* Prior exposure to TNF inhibitors including ETN. Prior exposure to efalizumab (Raptiva®) and alefacept (Amevive®) is also prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- South Korea (6):
  - Pfizer Investigational Site, Daejeon, Korea
  - Pfizer Investigational Site, Gyeonggido, Korea
  - Pfizer Investigational Site, Seoul, Korea
  - Pfizer Investigational Site, S0, Seoul
  - Pfizer Investigational Site, Seoul, Seoul
  - Pfizer Investigational Site, Seoul

REFERENCES:
- [Derived] Lee JH, Youn JI, Kim TY, Choi JH, Park CJ, Choe YB, Song HJ, Kim NI, Kim KJ, Lee JH, Yoo HJ. A multicenter, randomized, open-label pilot trial assessing the efficacy and safety of etanercept 50 mg twice weekly followed by etanercept 25 mg twice weekly, the combination of etanercept 25 mg twice weekly and acitretin, and acitretin alone in patients with moderate to severe psoriasis. BMC Dermatol. 2016 Jul 25;16(1):11. doi: 10.1186/s12895-016-0048-z. PMID 27455955
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A6-4625&StudyName=Study%20Evaluating%20the%20Efficacy%20and%20Safety%20of%20Etanercept%20and%20Acitretin%20in%20Korean%20Patient%20With%20Moderate%20to%20Severe%20Psoriasis%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Etanercept 50 milligram (mg) subcutaneous injection twice weekly (BIW) for 12 weeks followed by Etanercept 25 mg BIW for 12 weeks
- Etanercept and Acitretin: Etanercept 25 mg subcutaneous injection BIW and acitretin 10 mg twice per day (BID) for 24 weeks.
- Acitretin: Acitretin 10 mg subcutaneous injection BID for 24 weeks
Period: Overall Study
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Started | 21 | 20 | 19
Received Treatment | 21 | 20 | 18
Study Assessments Performed | 21 | 19 | 18
Completed | 17 | 16 | 12
Not Completed | 4 | 4 | 7
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin | Total
Number analyzed (Participants) | 21 | 19 | 18 | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 38.57 (9.53) | 35.5 (8.75) | 42.39 (11.95) | 38.78 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 3 | 10
  Male | 16 | 17 | 15 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a 75 Percent (%) Improvement in Psoriasis Area and Severity Index (PASI 75) Score at Week 24
Description: Combined assessment of lesion severity and area affected into single score; range: 0 (no disease) to 72 (maximal disease). Body was divided into 4 sections (head, arms, trunk, legs); each area scored by itself and scores combined for final PASI. For each section, area of skin involved was estimated: 0 (0%) to 6 (90 - 100%), and severity estimated by clinical signs: erythema, induration, and desquamation; scale: 0 (none) to 4 (exceptionally striking). Final PASI = sum of severity parameters for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
Time Frame: Week 24
Population: Modified intent to treat (mITT) population: randomized participants who took at least 1 dose of test article and had both baseline and on-therapy PASI evaluations; Last Observation Carried Forward (LOCF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
percentage of participants | 52.38 [29.78 to 74.29] | 57.89 [33.50 to 79.75] | 22.22 [6.41 to 47.64]
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference; Test type: Superiority or Other; p = 0.0672, Fisher Exact

2. Secondary Outcome: Percentage of Participants Achieving a 50% Improvement in Psoriasis Area and Severity Index (PASI 50) Score
Description: as for outcome 1
Time Frame: Weeks 2, 4, 8, 12, 18, and 24
Population: mITT; LOCF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
percentage of participants
  Week 2 | 4.76 [0.12 to 23.82] | 0 [0 to 0] | 0 [0 to 0]
  Week 4 | 47.62 [25.71 to 70.22] | 15.79 [3.38 to 39.58] | 11.11 [1.38 to 34.71]
  Week 8 | 71.43 [47.82 to 88.72] | 57.89 [33.50 to 79.75] | 27.78 [9.69 to 53.48]
  Week 12 | 76.19 [52.83 to 91.78] | 78.95 [54.43 to 93.95] | 22.22 [6.41 to 47.64]
  Week 18 | 76.19 [52.83 to 91.78] | 84.21 [60.42 to 96.62] | 38.89 [17.30 to 64.25]
  Week 24 | 71.43 [47.82 to 88.72] | 84.21 [60.42 to 96.62] | 44.44 [21.53 to 69.24]
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference Week 2; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference Week 4; Test type: Superiority or Other; p = 0.0229, Fisher Exact
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference Week 8; Test type: Superiority or Other; p = 0.0256, Fisher Exact
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference Week 12; Test type: Superiority or Other; p = 0.0004, Fisher Exact
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference Week 18; Test type: Superiority or Other; p = 0.0105, Fisher Exact
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference Week 24; Test type: Superiority or Other; p = 0.0366, Fisher Exact

3. Secondary Outcome: Percentage of Participants Achieving a Status on the Physician Global Assessment (PGA) of Psoriasis of Clear
Description: PGA of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease. Assessment of clear = PGA score of 0 (no evidence).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Percentage of participants
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Week 2 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Week 4 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Week 8 | 4.76 [0.12 to 23.82] | 0 [0 to 0] | 0 [0 to 0]
  Week 12 | 9.52 [1.17 to 30.38] | 0 [0 to 0] | 0 [0 to 0]
  Week 18 | 9.52 [1.17 to 30.38] | 5.26 [0.13 to 26.03] | 5.56 [0.14 to 27.29]
  Week 24 | 9.52 [1.17 to 30.38] | 10.53 [1.30 to 33.14] | 5.56 [0.14 to 27.29]
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.3230, Fisher Exact
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 1.0000, Fisher Exact

4. Secondary Outcome: Percentage of Participants Achieving a Status on the PGA of Psoriasis of Clear or Almost Clear
Description: PGA of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease. Assessment of clear or almost clear = PGA score of 0 (no evidence), or 1 (minimal/faint).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
percentage of participants
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Week 2 | 0 [0 to 0] | 0 [0 to 0] | 5.56 [0.14 to 27.29]
  Week 4 | 19.05 [5.45 to 41.91] | 5.26 [0.13 to 26.03] | 11.11 [1.38 to 34.71]
  Week 8 | 28.57 [11.28 to 52.18] | 21.05 [6.05 to 45.57] | 5.56 [0.14 to 27.29]
  Week 12 | 42.86 [21.82 to 65.98] | 21.05 [6.05 to 45.57] | 5.56 [0.14 to 27.29]
  Week 18 | 33.33 [14.59 to 56.97] | 31.58 [12.58 to 56.55] | 16.67 [3.58 to 41.42]
  Week 24 | 52.38 [29.78 to 74.29] | 52.63 [28.86 to 75.55] | 16.67 [3.58 to 41.42]
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.3103, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.4763, Fisher Exact
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.1961, Fisher Exact
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0272, Fisher Exact
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.5038, Fisher Exact
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0374, Fisher Exact

5. Secondary Outcome: Percentage of Participants Achieving a Status on the PGA of Psoriasis of Clear or Almost Clear or Mild
Description: PGA of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease. Assessment of clear or almost clear or mild = PGA score of 0 (no evidence), 1 (minimal/faint), 2 (mild).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
percentage of participants
  Baseline | 14.29 [3.05 to 36.34] | 5.26 [0.13 to 26.03] | 16.67 [3.58 to 41.42]
  Week 2 | 33.33 [14.59 to 56.97] | 26.32 [9.15 to 51.20] | 11.11 [1.38 to 34.71]
  Week 4 | 42.86 [21.82 to 65.98] | 47.37 [24.45 to 74.14] | 16.67 [3.58 to 41.42]
  Week 8 | 61.90 [38.44 to 81.89] | 42.11 [20.25 to 66.50] | 27.78 [9.69 to 53.48]
  Week 12 | 76.19 [52.83 to 91.78] | 78.95 [54.43 to 93.95] | 33.33 [13.34 to 59.01]
  Week 18 | 80.95 [58.09 to 94.55] | 84.21 [60.42 to 96.62] | 38.89 [17.30 to 64.25]
  Week 24 | 76.19 [52.83 to 91.78] | 84.21 [60.42 to 96.62] | 33.33 [13.34 to 59.01]
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Baseline; Test type: Superiority or Other; p = 0.6061, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.2971, Fisher Exact
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.1119, Fisher Exact
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.1081, Fisher Exact
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0063, Fisher Exact
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0055, Fisher Exact
Statistical Analysis 7: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0031, Fisher Exact

6. Secondary Outcome: Time to Achieve a PASI 50 Score
Description: PASI 50 defined as a 50% or greater improvement in PASI score from Baseline
Time Frame: Baseline up to Week 24
Population: mITT
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
days | 56 [28 to 56] | 56 [54 to 84] | 126 [56 to NA] — Not Available (NA): The number of events to observe the upper limit of 95% Confidence Interval (CI) did not occur during the specified period.
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference; Test type: Superiority or Other; p = 0.0033, Log Rank

7. Secondary Outcome: Time to Achieve a PASI 75 Score
Description: PASI 75 defined as a 75% or greater improvement in PASI score from Baseline
Time Frame: Baseline up to Week 24
Population: mITT
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
days | 126 [56 to 146] | 146 [124 to NA] — The number of events to observe the upper limit of 95% CI did not occur during the specified period. | NA [127 to NA] — The number of events to observe the median time to PASI 75 did not occur during the specified period.
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference; Test type: Superiority or Other; p = 0.0448, Log Rank

8. Secondary Outcome: Time to Achieve a Status on the PGA of Psoriasis of Clear or Almost Clear or Mild
Description: PGA of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease. Assessment of clear or almost clear or mild = PGA score of 0 (no evidence), 1 (minimal/faint), or 2 (mild).
Time Frame: Baseline up to Week 24
Population: mITT
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
days | 57 [19 to 84] | 57 [14 to 84] | 169 [56 to NA] — The number of events to observe the upper limit of 95% CI did not occur during the specified period.
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference; Test type: Superiority or Other; p = 0.0041, Log Rank

9. Secondary Outcome: Time to Achieve a Status on the PGA of Psoriasis of Clear or Almost Clear
Description: as for outcome 4
Time Frame: Baseline up to Week 24
Population: mITT
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
days | 167 [55 to 172] | 165 [59 to NA] — The number of events to observe the upper limit of 95% CI did not occur during the specified period. | NA [87 to NA] — The number of events to observe the median time to achieve PGA of Clear or Almost Clear did not occur during the specified period.
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference; Test type: Superiority or Other; p = 0.3536, Log Rank

10. Secondary Outcome: Change From Baseline in the PGA of Psoriasis
Description: PGA of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease. Assessment of clear = PGA score of 0 (no evidence). Change = Week x, minus Baseline, where smaller scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18, and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
units on a scale
  Baseline | 3.40 (0.82) | 3.38 (0.59) | 3.50 (0.92)
  Change at Week 2 | -0.51 (0.71) | -0.35 (0.58) | 0.02 (0.56)
  Change at Week 4 | -1.00 (1.03) | -0.84 (0.60) | -0.26 (0.74)
  Change at Week 8 | -1.34 (1.07) | -1.09 (0.86) | -0.43 (0.91)
  Change at Week 12 | -1.62 (1.33) | -1.42 (0.69) | -0.48 (0.98)
  Change at Week 18 | -1.58 (1.33) | -1.68 (1.00) | -0.69 (1.35)
  Change at Week 24 | -1.67 (1.47) | -1.86 (1.06) | -0.71 (1.37)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0203, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0102, ANCOVA
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0056, ANCOVA
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0006, ANCOVA
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0066, ANCOVA
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0058, ANCOVA

11. Secondary Outcome: Change From Baseline in the PASI Score
Description: Combined assessment of lesion severity, area affected into single score; range:0(no disease) to 72(maximal disease).Body divided into 4 sections (head, arms, trunk, legs); each area scored by itself and scores combined for final PASI. For each section, area of skin involved was estimated:0(0%) to 6(90-100%), severity estimated by clinical signs: erythema, induration, desquamation; scale: 0(none) to 4(maximum). Final PASI = sum of severity parameters for each section * area score * weight of section(head:0.1,arm:0.2,body: 0.3, leg:0.4). Change=Week X-Baseline, smaller scores show improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
units on a scale
  Baseline | 20.83 (14.02) | 19.75 (9.85) | 26.31 (13.63)
  Change at Week 2 | -5.38 (7.13) | -3.27 (1.88) | -3.17 (5.60)
  Change at Week 4 | -9.98 (10.64) | -6.45 (3.19) | -4.06 (5.68)
  Change at Week 8 | -11.11 (10.89) | -9.96 (3.73) | -6.84 (9.57)
  Change at Week 12 | -11.97 (11.63) | -11.39 (4.72) | -6.71 (6.81)
  Change at Week 18 | -12.13 (11.67) | -13.54 (6.80) | -8.77 (8.54)
  Change at Week 24 | -12.16 (12.15) | -13.92 (5.75) | -9.62 (10.10)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0329, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0003, ANCOVA
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0598, ANCOVA
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0241, ANCOVA
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0543, ANCOVA
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.1205, ANCOVA

12. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Involvement of Psoriasis at Weeks 2, 4, 8, 12, 18 and 24
Description: Change from Baseline in the percentage of the surface area of the body affected by psoriasis. Change = Week x minus Baseline, where smaller scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
percentage of BSA
  Baseline | 32.98 (20.21) | 32.50 (24.15) | 39.75 (22.96)
  Change at Week 2 | -2.64 (6.69) | -1.55 (5.07) | -0.36 (5.54)
  Change at Week 4 | -7.36 (10.89) | -4.50 (6.48) | -0.75 (7.66)
  Change at Week 8 | -12.67 (13.17) | -7.97 (9.27) | -5.14 (16.96)
  Change at Week 12 | -15.43 (14.90) | -10.29 (9.19) | -5.08 (11.89)
  Change at Week 18 | -16.57 (14.70) | -14.76 (11.61) | -9.25 (16.72)
  Change at Week 24 | -17.52 (14.91) | -16.87 (10.79) | -10.30 (18.86)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.1385, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0019, ANCOVA
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0442, ANCOVA
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0034, ANCOVA
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0454, ANCOVA
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0539, ANCOVA

13. Secondary Outcome: Change From Baseline in Subject Global Assessment (SGA) of Joint Pain at Weeks 2, 4, 8, 12 ,18 and 24
Description: Participants were asked to rate the severity of their joint pain on a 6-point scale, where 0=good and 5=severe. Change = Week X minus Baseline, where smaller scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF; Number of participants analyzed (N)= participants with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 18 | 18
units on a scale
  Baseline | 0.67 (1.43) | 0.56 (1.15) | 0.94 (1.73)
  Change at Week 2 | 0.00 (0.71) | 0.00 (0.49) | -0.44 (1.10)
  Change at Week 4 | 0.29 (1.19) | -0.06 (0.42) | -0.72 (1.81)
  Change at Week 8 | 0.19 (0.81) | -0.22 (0.88) | -0.56 (1.72)
  Change at Week 12 | 0.00 (0.63) | -0.28 (0.96) | -0.44 (2.36)
  Change at Week 18 | -0.05 (0.67) | -0.28 (1.02) | -0.44 (1.85)
  Change at Week 24 | 0.29 (1.06) | -0.39 (0.85) | -0.61 (2.03)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.1723, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0292, ANCOVA
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0908, ANCOVA
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.5678, ANCOVA
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.4820, ANCOVA
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0394, ANCOVA

14. Secondary Outcome: Change From Baseline in SGA of Psoriasis at Weeks 2, 4, 8, 12 ,18 and 24
Description: Participants were asked to rate the severity of their psoriasis disease activity on a 6-point scale, where 0=good and 5=severe. Change = Week X minus Baseline, where smaller scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12 ,18 and 24
Population: mITT; LOCF; Number of participants analyzed (N)= participants with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 18 | 18
units on a scale
  Baseline | 3.90 (1.09) | 3.94 (1.06) | 4.72 (0.67)
  Change at Week 2 | -0.90 (1.58) | -0.33 (1.24) | -0.72 (1.02)
  Change at Week 4 | -1.86 (1.28) | -0.94 (1.26) | -0.83 (1.04)
  Change at Week 8 | -2.29 (1.79) | -1.89 (1.49) | -1.67 (1.71)
  Change at Week 12 | -2.67 (1.56) | -2.28 (1.53) | -1.61 (1.72)
  Change at Week 18 | -2.57 (1.99) | -2.11 (1.78) | -1.83 (1.76)
  Change at Week 24 | -1.81 (2.20) | -2.39 (1.54) | -1.72 (1.93)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.1079, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0004, ANCOVA
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0146, ANCOVA
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0019, ANCOVA
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0062, ANCOVA
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0197, ANCOVA

15. Secondary Outcome: Change From Baseline in SGA of Itching at Each Visit
Description: Participants were asked to rate the severity of their psoriasis itching on a 6-point scale, where 0=good and 5=severe. Change = Week X minus Baseline, where smaller scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12 ,18 and 24
Population: mITT; LOCF; Number of participants analyzed (N)= participants with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 18 | 18
units on a scale
  Baseline | 3.33 (1.35) | 3.11 (1.81) | 3.72 (1.45)
  Change at Week 2 | -0.67 (1.59) | 0.28 (1.74) | -0.39 (1.29)
  Change at Week 4 | -1.52 (1.33) | -0.61 (1.65) | -0.39 (2.03)
  Change at Week 8 | -1.86 (2.06) | -1.06 (1.76) | -1.28 (1.71)
  Change at Week 12 | -2.10 (2.07) | -1.44 (2.09) | -1.22 (1.73)
  Change at Week 18 | -1.81 (2.06) | -1.83 (1.76) | -1.17 (1.62)
  Change at Week 24 | -1.19 (2.23) | -1.83 (2.04) | -1.06 (1.89)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.1229, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0136, ANCOVA
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.1578, ANCOVA
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0565, ANCOVA
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0685, ANCOVA
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0493, ANCOVA

16. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 1, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the overall appearance of their skin. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 0.67 (0.80) | 0.74 (0.99) | 0.44 (0.78)
  Change at Week 2 | 0.81 (1.25) | 0.79 (1.40) | 0.28 (1.41)
  Change at Week 4 | 1.57 (1.16) | 0.95 (1.31) | 0.50 (1.38)
  Change at Week 8 | 2.10 (1.58) | 1.58 (1.71) | 0.78 (1.40)
  Change at Week 12 | 2.10 (1.58) | 1.74 (1.76) | 0.56 (1.38)
  Change at Week 18 | 2.24 (1.87) | 1.95 (1.54) | 1.06 (1.66)
  Change at Week 24 | 1.76 (1.67) | 2.05 (1.18) | 1.11 (1.84)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.3112, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0196, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0109, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0035, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0603, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.2184, Kruskal-Wallis

17. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 2, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on the flaking of their skin. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 1.00 (1.30) | 0.84 (1.21) | 0.56 (0.78)
  Change at Week 2 | 1.14 (1.53) | 1.21 (1.51) | 0.39 (1.50)
  Change at Week 4 | 1.57 (1.36) | 0.68 (1.42) | 0.94 (1.66)
  Change at Week 8 | 2.38 (1.83) | 1.53 (1.95) | 1.11 (1.78)
  Change at Week 12 | 2.67 (1.88) | 1.63 (1.46) | 0.83 (1.76)
  Change at Week 18 | 2.33 (2.01) | 1.89 (1.41) | 1.28 (1.84)
  Change at Week 24 | 1.90 (2.17) | 2.21 (1.18) | 1.17 (1.86)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.1774, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.1195, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0606, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0030, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.1567, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.2094, Kruskal-Wallis

18. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 3, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on the redness of their skin. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 0.90 (1.18) | 0.63 (1.01) | 0.72 (0.89)
  Change at Week 2 | 0.86 (1.20) | 1.32 (1.34) | 0.17 (1.20)
  Change at Week 4 | 0.95 (1.24) | 1.16 (1.17) | 0.44 (1.04)
  Change at Week 8 | 2.05 (2.04) | 1.58 (1.71) | 0.83 (1.34)
  Change at Week 12 | 2.19 (1.97) | 1.68 (1.67) | 0.61 (1.38)
  Change at Week 18 | 2.05 (2.20) | 2.16 (1.21) | 1.22 (1.52)
  Change at Week 24 | 2.00 (2.02) | 2.21 (1.23) | 1.00 (1.41)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0302, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0980, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0711, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0077, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.1553, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0410, Kruskal-Wallis

19. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 4, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on tightness in the skin. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 1.33 (1.28) | 1.11 (1.05) | 1.83 (1.76)
  Change at Week 2 | 1.48 (1.50) | 0.42 (1.61) | -0.11 (1.57)
  Change at Week 4 | 2.19 (1.72) | 0.79 (1.13) | 0.44 (1.79)
  Change at Week 8 | 2.43 (2.34) | 1.32 (1.29) | 0.83 (1.76)
  Change at Week 12 | 2.67 (2.18) | 1.74 (1.48) | 0.61 (2.20)
  Change at Week 18 | 2.48 (2.16) | 2.05 (1.18) | 0.78 (1.77)
  Change at Week 24 | 1.90 (2.47) | 2.00 (1.05) | 0.56 (1.62)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0060, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0058, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0127, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0068, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0096, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0132, Kruskal-Wallis

20. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 5, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on bleeding of the skin. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 2.81 (1.86) | 2.84 (1.64) | 2.89 (2.14)
  Change at Week 2 | 0.57 (1.60) | 0.68 (1.53) | 0.28 (1.74)
  Change at Week 4 | 1.00 (1.95) | 0.74 (1.45) | 0.56 (2.09)
  Change at Week 8 | 1.43 (1.99) | 1.05 (1.22) | 0.44 (1.82)
  Change at Week 12 | 1.43 (2.23) | 0.74 (1.28) | 0.78 (2.41)
  Change at Week 18 | 1.38 (2.25) | 1.16 (1.92) | 0.67 (2.09)
  Change at Week 24 | 1.00 (2.32) | 0.84 (1.64) | 0.61 (2.20)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.6904, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.7021, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.2199, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.5071, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.4765, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.8662, Kruskal-Wallis

21. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 6, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on burning sensation of the skin. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 2.81 (1.69) | 2.37 (1.86) | 2.28 (2.05)
  Change at Week 2 | 0.57 (1.57) | 0.37 (1.30) | -0.44 (1.65)
  Change at Week 4 | 0.76 (1.81) | 0.89 (1.49) | -0.06 (2.53)
  Change at Week 8 | 0.86 (1.98) | 1.37 (1.54) | 0.78 (1.90)
  Change at Week 12 | 1.14 (1.96) | 1.16 (1.86) | 0.56 (2.28)
  Change at Week 18 | 1.24 (1.92) | 1.58 (1.71) | 0.61 (2.33)
  Change at Week 24 | 0.67 (2.35) | 1.05 (1.72) | 0.44 (2.06)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.1144, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.4509, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.4350, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.6085, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.2582, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.5490, Kruskal-Wallis

22. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 7, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on skin pain. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 2.95 (1.63) | 2.21 (1.78) | 2.72 (2.11)
  Change at Week 2 | 0.48 (1.75) | 0.89 (1.59) | 0.28 (1.96)
  Change at Week 4 | 0.90 (1.76) | 1.00 (1.41) | 0.50 (2.26)
  Change at Week 8 | 1.24 (2.00) | 1.32 (1.45) | 0.89 (2.30)
  Change at Week 12 | 1.29 (2.05) | 1.32 (1.45) | 0.78 (2.73)
  Change at Week 18 | 1.10 (2.02) | 1.63 (1.71) | 1.00 (2.45)
  Change at Week 24 | 0.62 (2.27) | 1.37 (1.89) | 0.67 (2.14)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.3287, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.4149, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.3837, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.6777, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.4976, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.4189, Kruskal-Wallis

23. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 8, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on joint pain. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 4.43 (1.16) | 3.79 (1.40) | 4.17 (1.58)
  Change at Week 2 | -0.33 (1.11) | -0.05 (1.18) | 0.17 (0.99)
  Change at Week 4 | -0.52 (1.21) | 0.05 (0.91) | 0.22 (1.77)
  Change at Week 8 | -0.33 (1.20) | 0.21 (1.03) | 0.33 (1.53)
  Change at Week 12 | -0.29 (1.15) | 0.21 (1.18) | 0.00 (2.35)
  Change at Week 18 | -0.14 (0.85) | 0.37 (1.38) | -0.28 (1.60)
  Change at Week 24 | -0.57 (1.47) | 0.05 (1.22) | 0.17 (1.95)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.4760, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.4040, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.4753, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.5084, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.2293, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.3822, Kruskal-Wallis

24. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 9, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on their comfort level with their personal appearance. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 1.14 (1.56) | 0.79 (0.79) | 0.83 (1.10)
  Change at Week 2 | 0.43 (1.21) | 0.63 (1.46) | -0.11 (1.23)
  Change at Week 4 | 0.90 (1.64) | 1.05 (1.43) | -0.11 (1.23)
  Change at Week 8 | 1.48 (1.91) | 1.58 (1.61) | 0.44 (1.29)
  Change at Week 12 | 1.52 (2.18) | 1.89 (1.41) | 0.17 (1.34)
  Change at Week 18 | 1.90 (2.51) | 1.68 (1.29) | 0.72 (1.45)
  Change at Week 24 | 1.57 (2.29) | 2.21 (1.13) | 0.78 (1.44)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.2691, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0142, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0383, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0026, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0475, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0205, Kruskal-Wallis

25. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 10, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on their anxiety. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 2.29 (1.87) | 1.89 (1.73) | 2.22 (1.80)
  Change at Week 2 | 1.05 (1.66) | 0.63 (1.89) | -0.39 (1.54)
  Change at Week 4 | 1.24 (1.55) | 1.21 (1.84) | -0.61 (1.61)
  Change at Week 8 | 1.57 (1.91) | 1.47 (1.95) | 0.33 (2.06)
  Change at Week 12 | 1.52 (2.14) | 1.68 (1.73) | 0.22 (2.60)
  Change at Week 18 | 1.57 (2.01) | 1.53 (1.87) | 0.56 (2.15)
  Change at Week 24 | 1.24 (1.95) | 1.58 (1.68) | 0.67 (2.25)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0512, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0024, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0946, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0935, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.2073, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.3415, Kruskal-Wallis

26. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 11, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on their depression. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 2.43 (1.91) | 1.95 (1.72) | 2.33 (1.85)
  Change at Week 2 | 0.95 (1.32) | 1.11 (1.63) | -0.11 (1.18)
  Change at Week 4 | 1.33 (1.59) | 1.26 (1.97) | -0.22 (1.59)
  Change at Week 8 | 1.38 (1.83) | 1.47 (2.20) | 0.28 (1.41)
  Change at Week 12 | 1.71 (2.05) | 1.58 (1.64) | 0.17 (2.04)
  Change at Week 18 | 1.57 (2.09) | 1.47 (1.81) | 0.61 (1.58)
  Change at Week 24 | 1.19 (2.02) | 1.68 (1.70) | 0.67 (1.50)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0202, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0090, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0742, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0445, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.2211, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.1982, Kruskal-Wallis

27. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 12, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on their fatigue. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 2.95 (1.75) | 1.74 (1.52) | 2.78 (1.73)
  Change at Week 2 | 0.48 (1.86) | 0.89 (1.56) | -0.72 (1.99)
  Change at Week 4 | 0.29 (1.76) | 0.68 (1.80) | -0.56 (2.01)
  Change at Week 8 | 0.29 (1.82) | 0.95 (2.07) | -0.33 (2.35)
  Change at Week 12 | 0.48 (1.89) | 0.95 (1.72) | -0.89 (2.42)
  Change at Week 18 | 0.48 (1.89) | 1.37 (1.61) | -0.61 (2.06)
  Change at Week 24 | 0.24 (2.02) | 1.21 (2.20) | -0.67 (2.06)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0409, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.1450, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.2010, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0424, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0090, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0116, Kruskal-Wallis

28. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 13, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on how others responded to their personal appearance at work/school. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 2.29 (1.85) | 1.53 (1.02) | 1.83 (1.62)
  Change at Week 2 | 0.00 (1.67) | 0.53 (1.50) | -0.39 (1.58)
  Change at Week 4 | 1.05 (1.69) | 0.74 (1.05) | -0.33 (1.91)
  Change at Week 8 | 1.00 (1.73) | 1.11 (1.56) | -0.22 (1.77)
  Change at Week 12 | 0.95 (1.91) | 1.53 (1.43) | -0.33 (1.88)
  Change at Week 18 | 0.95 (1.86) | 1.42 (1.57) | 0.11 (2.14)
  Change at Week 24 | 0.95 (1.99) | 1.63 (1.46) | -0.11 (2.05)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.3355, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0341, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0899, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0062, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.1241, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0393, Kruskal-Wallis

29. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 14, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with the treatment's effect on how their skin affected social and leisure activities. Responses were based on a 5-point scale: Very dissatisfied (0), Dissatisfied (1), Neither satisfied nor dissatisfied (2), Satisfied (3), Very satisfied (4), Never had this problem (5). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 0.95 (1.02) | 0.89 (0.94) | 1.39 (1.50)
  Change at Week 2 | 0.57 (1.36) | 0.74 (1.41) | -0.06 (1.43)
  Change at Week 4 | 1.10 (1.64) | 0.89 (0.99) | 0.22 (1.73)
  Change at Week 8 | 1.76 (1.79) | 1.58 (1.61) | 0.28 (1.45)
  Change at Week 12 | 2.10 (2.02) | 1.89 (1.52) | -0.06 (1.70)
  Change at Week 18 | 1.90 (1.84) | 1.68 (1.70) | 0.50 (1.82)
  Change at Week 24 | 1.57 (2.09) | 1.95 (1.61) | 0.28 (2.08)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.3402, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.1184, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0104, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0010, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0250, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0410, Kruskal-Wallis

30. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 15, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with their psoriasis therapy in general. Responses were based on a 5-point scale: very dissatisfied (0), dissatisfied (1), neither satisfied nor dissatisfied (2), satisfied (3), very satisfied (4). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 1.19 (1.12) | 1.37 (1.21) | 1.41 (1.18)
  Change at Week 2 | 1.24 (1.18) | 1.00 (1.60) | 0.18 (1.55)
  Change at Week 4 | 1.67 (1.20) | 1.00 (1.37) | 0.12 (1.58)
  Change at Week 8 | 1.67 (1.32) | 1.37 (1.83) | 0.53 (1.55)
  Change at Week 12 | 1.90 (1.51) | 1.53 (1.74) | 0.35 (1.87)
  Change at Week 18 | 1.86 (1.56) | 1.74 (1.52) | 0.82 (1.78)
  Change at Week 24 | 1.38 (1.47) | 1.68 (1.60) | 0.76 (1.95)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0894, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0084, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.0727, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0337, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.1380, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.3415, Kruskal-Wallis

31. Secondary Outcome: Change From Baseline in Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 16, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to respond to the statement "I would like to continue with my current psoriasis treatment". Responses were based on a 5-point scale: strongly disagree (0), disagree(1), neither agree nor disagree (2), agree (3), strongly agree (4). Change = Week X minus Baseline, where larger scores indicate improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Units on a scale
  Baseline | 3.10 (1.22) | 3.42 (1.02) | 2.82 (1.42)
  Change at Week 2 | 0.48 (1.17) | 0.11 (1.20) | 0.00 (1.80)
  Change at Week 4 | 0.67 (1.24) | 0.05 (1.18) | -0.12 (1.93)
  Change at Week 8 | 0.52 (1.54) | 0.26 (1.05) | 0.06 (1.98)
  Change at Week 12 | 0.48 (1.50) | 0.16 (1.21) | -0.29 (2.14)
  Change at Week 18 | 0.48 (1.50) | 0.21 (1.13) | -0.29 (2.08)
  Change at Week 24 | 0.14 (1.53) | 0.11 (1.10) | -0.18 (1.88)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.4407, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.1768, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.4636, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.3340, Kruskal-Wallis
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.1785, Kruskal-Wallis
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.7428, Kruskal-Wallis

32. Secondary Outcome: Change From Baseline in the Percentage of Participants Who Responded "Yes" to the Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 17, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to answer the following question with either a "yes" or "no", "Taking into account your psoriasis symptoms, the appearance of your skin and all other problems which psoriasis causes, do you consider that your current health state is satisfactory?" Percentage of participants who responded "yes" reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
Percentage of participants
  Baseline | 9.52 [1.17 to 30.38] | 15.79 [3.38 to 39.58] | 22.22 [6.41 to 47.64]
  Week 2 | 14.29 [3.05 to 36.34] | 42.11 [20.25 to 66.50] | 27.78 [9.69 to 53.48]
  Week 4 | 42.86 [21.82 to 65.98] | 52.63 [28.86 to 75.55] | 33.33 [13.34 to 59.01]
  Week 8 | 57.14 [34.02 to 78.18] | 57.89 [33.50 to 79.75] | 33.33 [13.34 to 59.01]
  Week 12 | 71.43 [47.82 to 88.72] | 57.89 [33.50 to 79.75] | 33.33 [13.34 to 59.01]
  Week 18 | 71.43 [47.82 to 88.72] | 63.16 [38.36 to 83.71] | 38.89 [17.30 to 64.25]
  Week 24 | 57.14 [34.02 to 78.18] | 73.68 [48.80 to 90.85] | 38.89 [17.30 to 64.25]
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Baseline; Test type: Superiority or Other; p = 0.5377, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.1419, Fisher Exact
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.5391, Fisher Exact
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.2589, Fisher Exact
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0635, Fisher Exact
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.1172, Fisher Exact
Statistical Analysis 7: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.1247, Fisher Exact

33. Secondary Outcome: Change From Baseline in the Percentage of Participants Who Responded "Yes" to Psoriasis Subject Satisfaction Questionnaire (PSSQ) Question 18, at Weeks 2, 4, 8, 12, 18 and 24
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to answer the following question with either a "yes" or "no", "Taking into account your psoriasis symptoms, the appearance of your skin, medicine side effects and medicine ease/difficulty of use, do you consider that your current psoriasis treatment is satisfactory?" Percentage of participants who responded "yes" reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 18 and 24
Population: mITT; LOCF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Number analyzed (Participants) | 21 | 19 | 18
percentage of participants
  Baseline | 38.10 [18.11 to 61.56] | 42.11 [20.25 to 66.50] | 33.33 [14.21 to 61.67]
  Week 2 | 80.95 [58.09 to 94.55] | 78.95 [54.43 to 93.95] | 50.00 [26.02 to 73.98]
  Week 4 | 85.71 [63.66 to 96.95] | 94.74 [73.97 to 99.87] | 55.56 [30.76 to 78.47]
  Week 8 | 90.48 [69.62 to 98.83] | 89.47 [66.86 to 98.70] | 66.67 [40.99 to 86.66]
  Week 12 | 95.24 [76.18 to 99.88] | 73.68 [48.80 to 90.85] | 61.11 [35.75 to 82.70]
  Week 18 | 90.48 [69.62 to 98.83] | 94.74 [73.97 to 99.87] | 61.11 [35.75 to 82.70]
  Week 24 | 80.95 [58.09 to 94.55] | 94.74 [73.97 to 99.87] | 55.56 [30.76 to 78.47]
Statistical Analysis 1: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Baseline; Test type: Superiority or Other; p = 0.9429, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 2; Test type: Superiority or Other; p = 0.0927, Fisher Exact
Statistical Analysis 3: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 4; Test type: Superiority or Other; p = 0.0151, Fisher Exact
Statistical Analysis 4: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 8; Test type: Superiority or Other; p = 0.1124, Fisher Exact
Statistical Analysis 5: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 12; Test type: Superiority or Other; p = 0.0242, Fisher Exact
Statistical Analysis 6: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 18; Test type: Superiority or Other; p = 0.0237, Fisher Exact
Statistical Analysis 7: Comparison: Etanercept vs Etanercept and Acitretin vs Acitretin; Overall treatment difference at Week 24; Test type: Superiority or Other; p = 0.0176, Fisher Exact

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept | Etanercept and Acitretin | Acitretin
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 1/18
Other Adverse Events (participants affected / at risk) | 14/21 | 14/20 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=21) | Etanercept and Acitretin (N=20) | Acitretin (N=18)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=21) | Etanercept and Acitretin (N=20) | Acitretin (N=18)
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 3 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 2
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Condition aggravated (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
One of the protocol-defined endpoints was change from baseline in the participant's assessment of general health, however data was collected and analyzed for change from baseline in the participant's assessment of joint pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.